CLINICAL TRIAL: NCT03290547
Title: A Multi-Center Pilot Study of a Novel Multi-Wavelength Laser for Tattoo Removal
Brief Title: Pilot Study of Multi-wavelength Laser for Tattoo Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-15-EN10
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Tattoo Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- arm-1 (Other): Cutera enLighten laser treatments that allows the user to choose a wavelength between 640nm to 800nm.
  Interventions: Device: Cutera enLighten laser

INTERVENTIONS:
Device: Cutera enLighten laser — Subjects will receive laser treatments.

SUMMARY:
To evaluate the safety and efficacy of an investigational version of the Cutera enLighten laser that offers muliple wavelengths for tattoo removal.

DETAILED DESCRIPTION:
Currently, the enLighten laser offers two wavelengths: 532nm and 1064nm. The version of the laser under investigation allows the user to choose a wavelength between 640nm to 800nm.

This is a multi-center prospective, open-label, uncontrolled pilot study in up to 75 male or female subjects, age 18 to 65 years, who desire laser removal of a tattoo containing single or multi-color ink. Subjects will receive laser treatments and will be followed at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, 18 to 65 years of age (inclusive).
2. Fitzpatrick Skin Type I - VI (Appendix 3).
3. Target tattoo contains single or multi-color ink.
4. Subject must be able to read, understand and sign the Informed Consent Form.
5. Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
6. Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and/or every day for the duration of the study, including the follow-up period.
7. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
8. Agree to not undergo any other procedure(s) for tattoo removal during the study (as applicable).
9. Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant for the duration of the study.

   -

Exclusion Criteria:

1. Participation in a clinical trial of a drug or another device in the target area during the study..
2. Target tattoo contains only black ink.
3. History of allergic reaction to pigments following tattooing..
4. History of allergy to local anesthetics.
5. History of allergy to topical antibiotics.
6. History of malignant tumors in the target area.
7. Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
8. Pregnant and/or breastfeeding.
9. Having an infection, dermatitis or a rash in the treatment area.
10. Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
11. Suffering from coagulation disorders or taking prescription anticoagulation medications.
12. History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
13. History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
14. History of vitiligo, eczema, or psoriasis.
15. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
16. History of seizure disorders due to light.
17. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
18. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
19. History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
20. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
21. Systemic use of corticosteroid or isotretinoin within 6 months of study participation.
22. Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
23. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
24. Current smoker or history of smoking within 6 months of study participation.
25. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, M.D., Principal Investigator — Cutera Research Center; Jeffrey Dover, M.D., Principal Investigator — Skin Care Physicians
Locations (2):
- United States (2):
  - Cutera Research Center, Brisbane, California
  - Skin Care Physicians, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cutera enLighten Laser: Cutera enLighten laser treatments that allows the user to choose a wavelength between 640nm to 800nm.
Period: Overall Study
Arm/Group | Cutera enLighten Laser
Started | 22
Completed | 6
Not Completed | 16

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: Cutera enLighten laser treatments that allows the user to choose a wavelength between 640nm to 800nm.
  Cutera enLighten laser: Subjects will receive up to 10 laser treatments.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Degree of Tattoo Clearing at 6 Weeks Post-final Treatment as Assessed by the Investigator
Description: Degree of tattoo clearing using the GAIS (Global Assessment of Improvement Scale) 3 = Very Significant Improvement, 2 = Significant Improvement, 1 = Moderate Improvement, or 0 = Mild or No Improvement Higher scores indicate better outcomes
Time Frame: 6 weeks post-final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cutera enLighten Laser
Number analyzed (Participants) | 6
score on a scale | 2 (0.9)

ADVERSE EVENTS:
Time Frame: 12 weeks post final treatment, up to 15 months
Groups:
- All Enrolled Subjects: Cutera enLighten laser treatments that allows the user to choose a wavelength between 640nm to 800nm.
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Subjects (N=22)
Erythema (Skin and subcutaneous tissue disorders) | 21
Edema (Skin and subcutaneous tissue disorders) | 22
Frosting (Skin and subcutaneous tissue disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03290547/Prot_000.pdf